CLINICAL TRIAL: NCT05137561
Title: Comparison of Robotic-arm Assisted 68 Ga PSMA PET/CT Guided Prostate Biopsy Versus MR Directed TRUS Guided (Cognitive Fusion) Prostate Biopsy in PIRADS 4 and 5 Lesions: A Pilot Study to Assess Diagnostic Performance and Patient Safety
Brief Title: Robotic-arm Assisted 68 Ga PSMA PET/CT Guided Prostate Biopsy Versus MR Directed Cognitive Fusion TRUS Guided Prostate Biopsy (PROBIOP)
Acronym: PROBIOP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajender Kumar, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NK/7840/MD/624
Record Dates: First submitted 2021-10-26; First posted 2021-11-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Simple randomization using RRApp
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSMA PET/CT guided biopsy arm (Active Comparator): PSMA PET/CT guided biopsy will be done from PSMA avid lesion of the prostate after reviewing the whole body PSMA PET/CT scan.
  Interventions: Procedure: PSMA PET guided prostate biopsy
- MRI directed TRUS guided biopsy (Active Comparator): The MRI-directed transrectal ultrasound-guided per-rectal prostate biopsy will be done by cognitive fusion.
  Interventions: Procedure: MRI directed TRUS guided prostate biopsy

INTERVENTIONS:
Procedure: PSMA PET guided prostate biopsy — PSMA PET-guided prostate biopsy from PSMA avid prostatic lesion will be done.
  Arms: PSMA PET/CT guided biopsy arm
Procedure: MRI directed TRUS guided prostate biopsy — TRUS guided MR directed Cognitive fusion prostate biopsy based on the PIRADS scoring
  Arms: MRI directed TRUS guided biopsy

SUMMARY:
The present study aimed to compare the diagnostic accuracy, radiation exposure, complication rates between 68Ga-PSMA PET/CT guided robotic arm assisted prostate biopsy and MRI directed TRUS guided prostate biopsy in PIRADS 4/5 lesions.

DETAILED DESCRIPTION:
To compare the diagnostic yield of Robotic-arm assisted 68Ga PSMA PET/CT guided prostate biopsy and MRI directed TRUS guided prostate biopsy in patients with PIRADS grading 4/5.

To compare the visual pain index of the patients between two arms during the procedure.

To compare the complication rates between the two arms during and after the procedure for a period of 2 weeks

ELIGIBILITY:
Inclusion Criteria:

1. PIRADS 4 and 5 prostate lesions and PIRADS </= 3 prostate lesions with high clinical suspicion.
2. Patients who are included in the study will be randomly allocated into either PSMA PET/CT guided biopsy or TRUS guided biopsy using simple randomization in RRApp

Exclusion Criteria:

1. Patients with acute prostatitis/ urine culture positive.
2. Patients with pre-existing bleeding diathesis like hemophilia, coagulopathy defined by INR ≥ 1.2, and Platelet counts ≤ 80,000/mm3
3. Patients who refuse to provide the written informed consent
4. Non-cooperative patients

Ages: 45 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is malignancy of the male prostate.
Enrollment: 217 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of mpMRI directed vs PET/CT directed prostate biopsy | 12 months
  The number of participants (with percentages) in whom the biopsy procedure yielded a tissue specimen adequate for a definite pathological diagnosis and detection of PCa in both arms
Diagnostic performance of mpMRI directed vs PET/CT directed prostate biopsy | 12 months
  The sensitivity, specificity and accuracy of mpMR directed TRUS guided (cognitive fusion) and PSMA PET/CT directed biopsy will be compared.

SECONDARY OUTCOMES:
Incidence of procedure related complications | three months
  The procedure-related complications in the number and percentage of recruiting participants will be tabulated.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol